CLINICAL TRIAL: NCT03543436
Title: Temocillin Versus a Carbapenem as Initial Intravenous Treatment for Extended-spectrum Beta-lactamase Related Urinary Tract Infections, a Non-inferiority Study
Brief Title: Temocillin Versus a Carbapenem as Initial Intravenous Treatment for ESBL Related Urinary Tract Infections
Acronym: TEMO-CARB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation Hôpital Saint-Joseph (Other); French National Network of Clinical Research in Infectious Diseases (RENARCI) (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 160910J; 2017-001257-14 (EudraCT Number)
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Urinary Tract Infections
Keywords: Non-inferiority study; Temocillin; Carbapenem; ESBL infection; Urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — temocillin; Meropenem; Imipenem; Carbapenems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous temocillin (Experimental): Intravenous temocillin 2g/intravenously/8h or renally adjusted equivalent (ORAE) in 30-40 min infusion or continuous intravenous (6g/24h)
  Interventions: Drug: Temocillin
- Intravenous meropenem or imipenem (Active Comparator): Intravenous meropenem or imipenem 1g/Intravenously /8h ORAE in 15-30 min infusion. Then switch to oral therapy
  Interventions: Drug: meropenem or imipenem

INTERVENTIONS:
Drug: Temocillin — Intravenous temocillin disodium 2g intravenously/8h Or Renally Adjusted Equivalent (ORAE) in 30-40 min infusion or continuous intravenous (6g/24h) .
  Arms: Intravenous temocillin
Drug: meropenem or imipenem — Intravenous carbapenem (meropenem 1g intravenously/8h Or Renally Adjusted Equivalent (ORAE) or imipenem 1g intravenously/8h ORAE)
  Other Names: Carbapenems
  Arms: Intravenous meropenem or imipenem

SUMMARY:
TEMO-CARB is a phase 3, randomized, controlled, multicentre, open-label pragmatic clinical trial to test the non-inferiority of temocillin versus carbapenem as initial intravenous treatment of Urinary Tract Infection (UTI) due to extended-spectrum beta-lactamase (ESBL) producing enterobacteriaceae.

DETAILED DESCRIPTION:
Urinary tract infections are among the most common bacterial infections that are treated in the community by an empirical antibiotic treatment regimen. Enterobacteriaceae are the most common bacteria involved in urinary tract infection. Since 2006, extended-spectrum beta-lactamase (ESBL) producing enterobacteriaceae have spread in France, as elsewhere. Finding therapeutic alternatives to carbapenems in infections caused by ESBL producing enterobacteriaceae is imperative. Although temocillin, 6-α-methoxy derivative of ticarcillin has been suggested as a potential alternative to carbapenem therapy for ESBL related infections, it was not investigated in accordance with current standard. The hypothesis to test in this study is that temocillin is not inferior to a carbapenem as initial intravenous treatment of urinary tract infections caused by ESBL producing enterobacteriaceae.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years)
* Hospitalized patient with clinically significant monomicrobial UTI
* Complicated UTI due to ESBL producing enterobacteriaceae (pyelonephritis, prostatitis or renal abscess) requiring parenteral antimicrobial therapy
* Susceptibility to temocillin and carbapenem as evidenced by testing results
* For woman able to procreate: negative pregnancy test and use of an effective method of contraception (abstinence, oral contraceptives, intra-uterine device, diaphragm with spermicide and condom). All forms of hormonal contraception are acceptable
* Signed informed consent by patient himself (able or under curatorship) or his legal representative (patient unable to give his consent or under tutorship)
* Patient affiliated to the social security system

Exclusion Criteria:

* Patient infected with a bacteria which is not an ESBL-producing enterobacteriaceae.
* Polymicrobial infection.
* Hypersensitivity and/or previous intolerance to carbapenem or temocillin, or penicillins or any other beta-lactam.
* Patient with a contraindication to any of the drugs to be used in research
* Patient presenting another site of infection than urinary (except onset of bacteraemia from urinary tract origin due to Gram negative bacteria).
* Woman who is pregnant, breastfeeding, or expecting to conceive at any time during the study (pregnancy test will be conducted for woman without menopause).
* Palliative care of life expectancy < 90 days.
* Ongoing empirical treatment of the urinary tract infections with carbapenem or temocillin > 24 hours before randomization
* Delay in randomization > 48 hours after identification of ESBL producing enterobacteriaceae in urinary and/or blood culture.
* Participation in other clinical trial for the infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Clinical and microbiological cure | 5-7 days after end of treatment
  The primary endpoint, was defined as achieving both clinical cure and microbiological eradication of all baseline pathogens 5-7 days after completion of treatment.
  Clinical cure is defined as complete resolution, substantial improvement or return to pre-infections signs and symptoms of complicated lower urinary tract infections or pyelonephritis without the need for additional antibiotic therapy Microbiological efficacy will be assessed by quantitative urine culture and defined as follows < 10^3 Colony Forming Unit (CFU)/mL of the baseline pathogens

SECONDARY OUTCOMES:
Early microbiological eradication | 3-4 days after randomization
  Microbiological eradication will be assessed by quantitative urine culture and defined as follows < 10^3 colony forming unit Colony Forming Unit (CFU)/mL of the baseline pathogens
Frequency of oral antibiotic switch in both arms (temocillin vs. carbapenem) | 60 days after randomization
Length of hospital stay | 60 days after randomization
  Time from randomization to hospital discharge
Persistent cure rate | 60 days after randomization
  Clinical cure is defined as complete resolution, substantial improvement or return to pre-infections signs and symptoms of complicated lower urinary tract infections or pyelonephritis without the need for additional antibiotic therapy
Clinical recurrences | 60 days after randomization
  Relapse: new symptoms of urinary tract infection in a patient previously considered as clinically or microbiologically cured in the visit 5-7 days after treatment completion plus positive urine ± blood culture grows the same microorganism isolated that in the initial culture.
  Re-infection: same definition but with different strain in urinary culture
Mortality | 60 days after randomization
  Death for any reason or for infectious events
Pharmacokinetic of temocillin according to kidney function | 3 days after treatment initiation
  Description of the temocillin plasma concentration and its variability among patients
Microbiota impact study | Time Frame : 5-7 days after treatment completion
  Study treatment impact in the gut colonization with multidrug Gram negative bacilli) and temocillin resistant Gram negative bacilli

CONTACTS AND LOCATIONS:
Overall Officials: Benoit PILMIS, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Olivier LORTHOLARY, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (16):
- France (16):
  - CHU de Martinique, Fort-de-france, Martinique
  - CHRU La Cavale Blanche, Brest
  - CHU de Grenoble Hospital, Grenoble
  - Melun Hospital - CHU Sud, Melun
  - APHP - Cochin Hospital, Paris
  - APHP - Necker-Enfants maladies Hospital, Paris
  - Bichat hospital, Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Tenon Hospital, Paris
  - APHP - Beaujon Hospital, Paris
  - APHP - Georges Pompidou European Hospital, Paris
  - APHP - Saint-Antoine Hospital, Paris
  - Saint-Joseph Hospital, Paris
  - CHU de Pau, Pau
  - CHU de Poitiers, Poitiers
  - CHU Pontchaillou, Rennes

IPD SHARING:
Plan to Share IPD: No